CLINICAL TRIAL: NCT05755568
Title: Characterization of Metachromatic Leukodystrophy (MLD) in Pediatric Population in Spain: Epidemiological, Clinical, Diagnostic, Therapeutic, and Socioeconomic Aspects
Brief Title: A Study to Learn About Metachromatic Leukodystrophy (MLD) in Children in Spain
Acronym: mECHromatic
Status: Withdrawn | Type: Observational
Why Stopped: Company decision after projects re-evaluation, taken before the study initiation.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-611-5002
Record Dates: First submitted 2023-02-02; First posted 2023-03-06 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Metachromatic Leukodystrophy (MLD)
Keywords: Drug Therapy
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MLD Participants: Data from medical records of participants diagnosed with late infantile or juvenile MLD at any time from 1 January 2000 to 31 December 2022 will be observed retrospectively.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this is an observational study, no intervention will be administered.

SUMMARY:
The main aim of this study is to learn about metachromatic leukodystrophy (MLD) in children and teenagers in Spain. This includes checking the number of new MLD cases and the frequency of children with MLD in 2022 in Spain.

There is no treatment involved in this study. Participants' data will be taken from their medical records (charts), which were already collected as a part of their routine care between 01 January 2000 and 31 December 2022.

DETAILED DESCRIPTION:
This is a non-interventional, retrospective study of participants diagnosed with late infantile or juvenile MLD whose data will be retrieved from existing health records.

Data from all participants, diagnosed with MLD from 01 January 2000 to 31 December 2022 will be collected from health records, including demographic and clinical data from the pre-diagnosis until the date of data collection or death, whatever occurs first.

The study will be conducted in Spain. The overall duration for data extraction is up to approximately 23 years.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosed with late infantile or juvenile MLD at any time between 01 January 2000 and 31 December 2022 (genetically and/or biochemically confirmed).

Exclusion Criteria:

• This study has no exclusion criteria.

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants diagnosed with late infantile or juvenile MLD in Spain.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Number of New Cases Diagnosed With MLD During Year 2022 | 1 year
  Data for Year 2022 will be considered as a part of retrospective data collection from 01 January 2000 to 31 December 2022 obtained from health records.
Number of New Cases Diagnosed With MLD per Subgroups of Phenotype During Year 2022 | 1 year
  Data for Year 2022 will be considered as a part of retrospective data collection from 01 January 2000 to 31 December 2022 obtained from health records.
Overall Number of Participants With MLD Alive On 31 December 2022 | 1 day
  Data for this outcome measure will be collected on last day of retrospective data collection from 01 January 2000 to 31 December 2022 obtained from health records.
Number of Participants With MLD Alive On 31 December 2022 per Subgroups of Phenotype | 1 day
  Data for this outcome measure will be collected on last day of retrospective data collection from 01 January 2000 to 31 December 2022 obtained from health records.
Overall Number of Participants With MLD Alive at Any Time During Year 2022 | 1 year
  Data for Year 2022 will be considered as a part of retrospective data collection from 01 January 2000 to 31 December 2022 obtained from health records.
Number of Participants With MLD Alive at Any Time During Year 2022 per Subgroups of Phenotype | 1 year
  Data for Year 2022 will be considered as a part of retrospective data collection from 01 January 2000 to 31 December 2022 obtained from health records.

SECONDARY OUTCOMES:
Number of Late Infantile and Juvenile (Early Juvenile and Late Juvenile) Phenotypes in Participants With MLD | 23 years
Age at Symptom Onset in Participants With MLD | 23 years
  Age at symptom onset in participants with MLD in years will be recorded.
Number of Participants With MLD Categorized Based on Clinical Signs/ Symptoms at Disease Onset | 23 years
  Clinical signs and symptoms include impaired gross motor skills, impaired fine motor skills, impaired language skills, impaired non-verbal communication, cognition, feeding/swallowing difficulties, skeletal deformity, musculoskeletal pain.
Age of Participants at Diagnosis of MLD | 23 years
  Age of participants at diagnosis of MLD in years will be recorded.
Time of Diagnosis Delay | 23 years
  Time of diagnosis delay will be computed as age at diagnosis minus age at symptom onset.
Number of Participants With Disease Diagnosis Based on Different Suggestive Findings | 23 years
  Suggestive findings will include motor, cognitive, behavioural, magnetic resonance imaging (MRI) and magnetic resonance (MR) spectroscopy.
Number of Participants With Disease Diagnosis Based on Confirmatory Tests | 23 years
  Confirmatory tests will include urine sulfatides, arylsulfatase A (ARSA) activity, ARSA genetic variants.
Number of Interactions of Participants With the Healthcare System Post Diagnosis | 1 year
  Interactions will include visits to nurses, rehabilitators, specialist, and other healthcare professionals (HCPs), attendance to emergency department, hospitalization, hospitalization days, surgery, and MLD-related procedures.
Number of Interactions of Participants With the Healthcare System Post Diagnosis Categorized by Type | 1 year
  Interactions will be categorized as: visits to nurses, rehabilitators, specialist, and other HCPs, attendance to emergency department, hospitalization, hospitalization days, surgery, and MLD-related procedures.
Number of Participants With Disease Progression | 23 years
  Disease progression will be analysed using brain MRI, MR spectroscopy, weight, height, and head circumference, fine motor function, gross motor function, speech function (expressive language), non-verbal communication, musculoskeletal symptoms, eating/drinking ability, cognitive status, social/behavioural function, nerve conduction and sleep quality.
Number of Treatment Types Used for MLD and Sequencing | 23 years
Percentage of Participants Under Specific MLD Treatments With Attenuated Disease Progression | 23 years
  The percentage of participants under specific MLD treatments with attenuated disease progression will be assessed using the participants' electronic medical records.
Number of Participants With Comorbidities and Complications | 23 years
Number of Participants With the Different Types of Symptomatic/Palliative Treatments and Supports | 23 years
Mortality Rate Based on Percentage of Participant-Deaths Per Year | 23 years
  Mortality rate is defined as proportion of deaths per year.
Proportion of Participant-Deaths Categorized by Cause of Death | 23 years
  Proportion of deaths categorized by cause of death will be recorded.
Age of Participants With MLD at Death | 23 years
  Age of MLD participants at death in years will be recorded.
Time From Onset of Symptoms to Death | 23 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- Spain (10):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruna
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario Vall dHebron, Barcelona
  - Hospital Universitario Infantil Nino Jesus, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No
Takeda does not provide access to Individual Participant Data when a study is in a very limited (small) study population due to participant privacy concerns such as potential reidentification of study participants.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/989b1eca0c2346e4?idFilter=%5B%22TAK-611-5002%22%5D